CLINICAL TRIAL: NCT05142709
Title: Real-world Experience of Anti-PD-1 Immunotherapy Plus Chemotherapy as First-line Treatment for Patients With Advanced Oesophageal Squamous Cell Carcinoma in China(REACTION Trial).
Brief Title: Real-world Experience of ICIs Plus Chemotherapy for Advanced ESCC.
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Other Study IDs: ESO-Shanghai18
Record Dates: First submitted 2021-10-31; First posted 2021-12-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESCC patients treated with anti-PD-1 immunotherapy as 1st line treatment.
  Interventions: Drug: Anti-PD-1 Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: Anti-PD-1 Immune Checkpoint Inhibitors — used as 1st line treatment for metastatic ESCC.

SUMMARY:
This study is a multi-center, non-interventional study. Clinicopathologic, treatment , outcome and efficacy data will be collected from medical records in metastatic esophageal squamous cell carcinoma (ESCC) patients.

DETAILED DESCRIPTION:
This study is a multi-center, non-interventional study. Patients' background, treatment pattern, treatment outcome, efficacy will be collected in metastatic esophageal squamous cell carcinoma (ESCC) patients who were treated with ICIs as 1st line treatment at approximately 26 institutions. The patients should have received at least 1 cycle of anti-PD-1 immunotherapy with or without radiotherapy. Based on these data, overall survival (OS), progression free survival (PFS) from start of 1st line treatment and the role and efficacy of radiotherapy for these patients will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Age > 18, had an Eastern Cooperative Oncology Group performance status score of 0-3; Patients had unresectable or recurrent disease that precluded esophagectomy or definitive chemoradiation, or distant metastatic disease; Patients had received no previous systemic therapy (patients who had progressed ≥6 months after [neo]adjuvant therapy or definitive chemoradiation were eligible); Patients accepted at least one cycle of anti-PD-1 immunotherapy as 1st line treatment, combined chemotherapy was allowed.

Patients who provided informed consent by appropriate methods. In dead case, optout will be applicable.

Exclusion Criteria:

Patients who are prior exposure to immune-mediated therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: More than 600 patients
Sampling Method: Non-Probability Sample
Enrollment: 1197 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
OS from start of 1st line treatment in metastatic ESCC | 2 years
  Median OS and OS rate at 12 months, 18 months and 24 months will be analysed based on Kaplan-Meier method and presented along with its 95% confidence interval.

SECONDARY OUTCOMES:
PFS from start of 1st line treatment in metastatic ESCC | 18 months
  Median PFS and PFS rate at 6 months, 12months and 18 months will be analysed based on Kaplan-Meier method and presented along with its 95% confidence interval.
the role of radiotherapy for patients treated with 1st immunotherapy. | 2 years
  Compare the median OS and PFS and the rates between the group of patients treated with or without radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lvhua Wang, M.D., Principal Investigator — Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center; Kuaile Zhao, M.D., Principal Investigator — Fudan University
Locations (23):
- China (23):
  - The 2nd affiliated hospital of Bengbu medical University, Bengbu, Anhui
  - The 2nd people's hospital of Anhui province, Hefei, Anhui
  - Fujian Cancer Hospital & Fujian Medical University Cancer Hospital, Fuzhou, Fujian
  - The 1st affiliated hospital of Xiamen University, Xiamen, Fujian
  - Cancer Hospital Chinese Academy of Medical Sciences,Shenzhen Center, Shenzhen, Guangdong
  - The 4th affiliated hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Anyang cancer hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan University Zhongnan hospital, Wuhan, Hubei
  - Zhongnan University Xiangya Hospital, Changsha, Hunan
  - Huai'an first hospital, Huai'an, Jiangsu
  - Jiangsu cancer Hosipital, Nanjing, Jiangsu
  - Nantong cancer hospital, Nantong, Jiangsu
  - Yancheng the 3rd hospital, Yancheng, Jiangsu
  - The Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The 1st affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The 2nd affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - Fudan University Shanghai cancer center, Shanghai, Shanghai Municipality
  - Sichuan cancer hospital, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The 2nd affiliated hospital of Wenzhou medical university, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No